CLINICAL TRIAL: NCT01044342
Title: A Single-centre, Randomised, Double-blind, Placebo-controlled, Four-period Cross-over Study to Evaluate the Scopolamine Cognition Model in Healthy Male Subjects Using AZD1446 and Donepezil Versus Placebo
Brief Title: A Healthy Volunteer Study to Evaluate Reversibility of Induced Impairment of Cognition
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: MSD, AstraZeneca
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: D2285M00021
Record Dates: First submitted 2010-01-06; First posted 2010-01-07 (Estimated); Last update posted 2010-05-10 (Estimated); Status verified 2010-05

CONDITIONS: Cognition
Keywords: Healthy Volunteers; EEG
MeSH Terms: interventions — 3-(5-chloro-2-furoyl)-3,7-diazabicyclo(3.3.0)octane; Donepezil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- A (Experimental): Single dose of AZD1446 10 mg
  Interventions: Drug: AZD1446
- B (Experimental): Single dose of AZD1446 80 mg
  Interventions: Drug: AZD1446
- C (Active Comparator): Single Dose of Donepezil 5 mg
  Interventions: Drug: donepezil
- D (Placebo Comparator): Single dose of placebo to match AZD1446
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD1446 — capsule; single oral dose
  Arms: A
Drug: AZD1446 — capsule, single oral dose
  Arms: B
Drug: donepezil — capsule, single oral dose
  Other Names: Aricept
  Arms: C
Drug: Placebo — capsule, single oral dose
  Arms: D

SUMMARY:
The purpose of this study is to determine if cognitive impairment induced by scopolamine is reversed using donepezil and/or AZD1446 as compared to placebo, as assessed by electroencephalogram (EEG) measures.

ELIGIBILITY:
Inclusion Criteria:

* BMI 18-30
* Non-smoker for at least 4 weeks

Exclusion Criteria:

* Any clinically relevant acute or chronic disease
* Hypersensitivity to scopolamine
* History of substance abuse

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2009-12; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
qEEG assessed through the absolutes alpha-power of the two occipital leads | In each treatment period (1, 2, 3, 4) the measure will be taken on Day 1 prior to dosing of AZD1446 or placebo and1h, 2h, 3h, 6h, and 24 hour after dosing of AZD1446 or placebo

SECONDARY OUTCOMES:
qEEGs/ERPs assessed by mismatch negativity and p300 | In each treatment period (1, 2, 3, 4) the measure will be taken on Day 1 prior to dosing of AZD1446 or placebo and1h, 2h, 3h, 6h, and 24 hour after dosing of AZD1446 or placebo

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Rouffach, France